CLINICAL TRIAL: NCT05208762
Title: A Phase 1 Study of PF-08046054/SGN-PDL1V in Advanced Solid Tumors
Brief Title: A Study of PF-08046054/SGN-PDL1V in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNPDL1V-001; C5851001 (Other: Alias Study Number); 2023-506604-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-12-15; First posted 2022-01-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of the Head and Neck; Esophageal Squamous Cell Carcinoma; Ovarian Neoplasms; Melanoma; Triple Negative Breast Neoplasms; Gastric Cancer
Keywords: Non-small cell lung cancer; NSCLC; Head and neck squamous cell carcinoma; HNSCC; Ovarian cancer; Triple Negative Breast Cancer; TNBC; Gastric cancer; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Ovarian Neoplasms; Melanoma; Triple Negative Breast Neoplasms; Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-08046054 Monotherapy (Experimental): PF-08046054 monotherapy
  Interventions: Drug: PF-08046054
- PF-08046054 Combination Therapy (Experimental): PF-08046054 + pembrolizumab
  Interventions: Drug: PF-08046054; Drug: pembrolizumab

INTERVENTIONS:
Drug: PF-08046054 — Given into the vein (IV; intravenously)
  Other Names: SGN-PDL1V
Drug: pembrolizumab — 200 mg once every 3 weeks given into the vein (IV; intravenously)
  Other Names: Keytruda
  Arms: PF-08046054 Combination Therapy

SUMMARY:
This study will test the safety of a drug called PF-08046054/SGN-PDL1V alone and with pembrolizumab in participants with solid tumors. It will also study the side effects of this drug. A side effect is anything a drug does to your body besides treating your disease.

Participants will have solid tumor cancer that has spread through the body (metastatic) or cannot be removed with surgery (unresectable).

This study will have five parts. Parts A and B of the study will find out how much PF-08046054/SGN- PDL1V should be given to participants. Part C will use the dose found in Parts A and B to find out how safe PF-08046054/SGN-PDL1V is and if it works to treat solid tumor cancers. In Part D and E, participants will be given PF-08046054/SGN-PDL1V with pembrolizumab to find out how safe this combination is and if it works to treat solid tumor cancers.

ELIGIBILITY:
Inclusion Criteria:

* Parts A and B:

  * Participants must have one of the following histologically- or cytologically-confirmed metastatic or unresectable solid tumor types

    * Non-small cell lung cancer (NSCLC)
    * Head and neck squamous cell carcinoma (HNSCC) (except nasopharyngeal cancer)
    * Esophageal squamous cell carcinoma (SCC)
    * Triple negative breast cancer (TNBC)
  * Participants must have disease that is relapsed or refractory, that has progressed on approved therapies, be intolerant to or refused such therapies, or such and therapies are contraindicated and in the judgement of the investigator, should have no appropriate SoC therapeutic option
  * Participants must have PD-L1 expression based on historical testing
* Part C:

  * Participants must have disease that is relapsed or refractory or be intolerant to SoC therapies and must have one of the following tumor types

    * HNSCC

      * Participants with HNSCC must have histologically or cytologically-confirmed HNSCC
    * NSCLC

      * Participants must have histologically or cytologically-confirmed NSCLC. Participants with SCC and non--SCC histology are eligible. Note: Participants with a neuroendocrine component or histology are not eligible.
    * Esophageal SCC
    * Ovarian cancer
    * Melanoma
    * TNBC
    * Gastric cancer
  * Participants must have been previously tested for PD-L1 expression and should have PD-L1 expression ≥1 or <1 by CPS or TPS based on historical testing
* Part D and Part E:

  * Participants must have histologically or cytologically-confirmed disease of the HNSCC or NSCLC
  * Participants must have PD-L1 expression based on historical testing
  * Participants with NSCLC; PD-L1 expression ≥ 1% by TPS
  * Participants with HNSCC; PD--L1 expression ≥1 by CPS
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Measurable disease per RECIST v1.1 at baseline

Exclusion Criteria:

* History of another malignancy within 3 years of first dose of study treatment or any evidence of residual disease from a previously diagnosed malignancy.
* Known active central nervous system metastases. Participants with previously-treated brain metastases may participate provided they:

  * Are clinically stable for at least 4 weeks prior to study entry after brain metastasis treatment
  * Have no new or enlarging brain metastases
  * And are off of corticosteroids prescribed for symptoms associate with brain metastases for at least 7 days prior to first dose of study treatment
* Lepto-meningeal disease
* Prior treatment with an anti-PD-L1 agent within less than 5 half-lives. This duration of time will vary according to the half-life of the specific agent.
* Previous receipt of an monomethylauristatin E (MMAE)-containing agent.
* Pre-existing neuropathy ≥Grade 2 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.

There are additional inclusion criteria. The study center will determine if criteria for participations are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2028-04-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through approximately 90 days after last study treatment; up to 3 years
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities | Through approximately 90 days after last study treatment; up to 3 years
Number of participants with dose-limiting toxicities (DLTs) | Through the first cycle of study treatment; approximately 1 month
Number of participants with DLTs by dose level | Through the first cycle of study treatment; approximately 1 month

SECONDARY OUTCOMES:
Confirmed objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) by investigator assessment | Up to approximately 3 years
  The proportion of participants with a partial response (PR) or complete response (CR) which is subsequently confirmed per RECIST v1.1 as assessed by the investigator.
Duration of objective response (DOR) per RECIST v1.1 by investigator assessment | Up to approximately 3 years
  The time from the start of the first documentation of objective tumor response (CR or PR that is subsequently confirmed) to the first documentation of PD (per RECIST v1.1 as assessed by the investigator) or to death due to any cause.
Progression-free survival (PFS) per RECIST v1.1 by investigator assessment | Up to approximately 3 years
  The time from the start of study treatment to the first documentation of PD (per RECIST v1.1 as assessed by the investigator) or death due to any cause.
Overall survival (OS) | Up to approximately 3 years
  The time from the start of study treatment to death due to any cause.
Pharmacokinetic (PK) parameter - Area under the concentration-time curve (AUC) | Through 30-37 days after last study treatment; up to approximately 3 years
  To be summarized using descriptive statistics
PK parameter - Maximum concentration (Cmax) | Through 30-37 days after last study treatment; up to approximately 3 years
  To be summarized using descriptive statistics
PK parameter - Trough concentration (Ctrough) | Through 30-37 days after last study treatment; up to approximately 3 years
  To be summarized using descriptive statistics
Incidence of anti-drug antibodies (ADAs) | Through 30-37 days after last study treatment; up to approximately 3 years
  To be summarized using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, IDS Pharmacy, Birmingham, Alabama
  - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, Davis Medical Center, Sacramento, California
  - The University of Iowa, Iowa City, Iowa
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Texas Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center - Redbird, Dallas, Texas
  - Univ. of TX Southwestern Medical Center - Zale Lipshy University Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center - William P. Clements, Jr., University Hospital, Dallas, Texas
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern - Simmons Cancer Center - Fort Worth, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center Investigational Pharmacy Services, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - UT Southwestern - Simmons Cancer Center - Richardson/Plano, Richardson, Texas
  - NEXT Virginia, LLC, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia
- Institut Jules Bordet, Anderlecht, Belgium
- Canada (3):
  - University Health Network, Toronto, Ontario
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (4):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
- France (5):
  - Hôpital Saint André - CHU Bordeaux, Bordeaux
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - lnstitut Curie Pharmacy, Paris
  - Institut Curie, Paris
  - Gustave Roussy Institute - Service pharmacie, Villejuif
- Germany (3):
  - Charite Comprehensive Cancer Center, Berlin
  - Charite Universitatsmedizin Berlin, Berlin
  - Apotheke-Zytostatika Studien Charite- Universitatsmedizin Berlin Campus Virchow Klinkum, Berlin
- Italy (4):
  - Divisione di Sviluppo di Nuovi Farmaci per Terapie Innovative lstituto Europeo di Oncologia, Milan, Milan
  - Centro Ricerche Cliniche di Verona s.r.l. c/o Policlinico G.B Rossi, Verona, Other
  - Azienda Ospedaliera Universitaria Integrata Verona - Policlinico G.B Rossi, Verona, Veneto
  - UOC Oncologia - IRCCS Azienda Ospedaliero Universitaria Bologna, Bologna
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
- The Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (6):
  - CETIR Viladomat, Barcelona, Other
  - Hospital Duran I Reynals-Institut Català d'Oncologia L'Hospitalet (ICO L'Hospitalet), Barcelona, Other
  - Hospital Quiron Salud Barcelona, Barcelona
  - NEXT Oncology Barcelona - IOB - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - START Madrid - CIOCC - Hospital Universitario HM Sanchinarro, Madrid
- United Kingdom (7):
  - Diagnostic Centre, London, Others
  - The Harley Street Clinic (THSC), London, Other
  - Pharmacy: Royal Marsden Hospital, Sutton, Surrey
  - Royal Marsden Hospital, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute, London
  - Radiology, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNPDL1V-001